CLINICAL TRIAL: NCT02799082
Title: A Randomized, Double-Blind, Phase III Multi-Center Study Evaluating the Safety and Efficacy of BF-200 ALA Versus Placebo in the Treatment of Actinic Keratosis (AK) When Using PDT
Brief Title: Evaluation of Efficacy and Safety of BF-200 ALA Used With Photodynamic Therapy in Patients With Actinic Keratosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biofrontera Bioscience GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALA-AK-CT003
Record Dates: First submitted 2016-05-27; First posted 2016-06-14 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — BF-200 ALA; Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Topical application of matched placebo gel (without containing active ingredient). Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1.0 cm surrounding margin.
  Interventions: Drug: Vehicle
- BF-200 ALA (Active Comparator): Topical application of BF-200 ALA gel containing 78 mg/g 5-aminolevulinic acid. Application of a 1 mm thick layer covering each lesion and a 0.5 cm to 1.0 cm surrounding margin.
  Interventions: Drug: BF-200 ALA

INTERVENTIONS:
Drug: Vehicle — topical treatment for photodynamic therapy combining vehicle application and subsequent illumination with broad or narrow spectrum light sources (after 3 h of drug incubation).
  Arms: Vehicle
Drug: BF-200 ALA — topical treatment for photodynamic therapy combining drug application and subsequent illumination with broad or narrow spectrum light sources (after 3 h of drug incubation).
  Other Names: Ameluz
  Arms: BF-200 ALA

SUMMARY:
The aim of the study was to evaluate the efficacy and safety of BF-200 ALA (Ameluz) used with photodynamic therapy (PDT) in patients suffering from actinic keratosis.

DETAILED DESCRIPTION:
The treatment comprised of one PDT session. If 12 weeks after PDT all lesions were cleared the patient entered the follow-up period. In case of remaining lesions or not completely cleared lesions the patient received a second PDT on the same day. The final assessment was performed 12 weeks after the last PDT and the patient moved to the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were willing and able to sign informed consent form.
* Men and women aged between 18 and 85 years inclusive.
* Subjects had a general good and stable health condition as confirmed by a physical examination and by medical history.
* Subjects with clinically stable medical conditions including, but not limited to the following diseases were allowed to be included into the study, if the medication taken for the treatment of the disease did not match the criteria of the excluded or disallowed medications listed in points 7, 10, 11 and 12 of the exclusion criteria:

  * controlled hypertension
  * diabetes mellitus type II
  * hypercholesterolemia
  * osteoarthritis
* Subjects accepted to abstain from sunbathing and the solarium during the study.
* Subjects had at least 4 but not more than 8 clinically confirmed actinic keratosis (AK) target lesions of mild to moderate intensity within the face or bald scalp (excluding eyelids, lips and mucosa), i.e. AK grade I and II according to Olsen et. al. 1991.
* To document and confirm the diagnosis of the investigators:

  * Photodocumentation of a representative lesion had to be evaluated and confirmed by an independent expert.
  * A pre-study biopsy had to be taken from a second representative AK lesion and was histopathologically evaluated by a dermato-pathological expert.
* If the evaluation of the photo by the independent reviewer could not confirm the diagnosis of the investigator, then the biopsy result decided whether the subject was eligible for the study.
* The AK lesions had to be discrete and quantifiable; the distance from one lesion to its neighbor lesion was greater than 1.0 cm
* The diameter of each AK lesion was not less than 0.5 cm and not greater than 1.5 cm. The size of each baseline AK lesion was recorded by measuring the two largest perpendicular diameters. To describe irregular lesions (ellipsoidal) investigators measured the major and minor axis. Both axes had to be above the minimum of 0.5 cm and less than 1.5 cm.
* The subjects were free of any significant physical abnormalities (e.g., tattoos, dermatoses) in the potential treatment area that might cause difficulty with examination or final evaluation.
* The subjects were willing to stop using moisturizers and any other topical treatments with anti-aging products, vitamin A, vitamin C, and/or vitamin E containing ointments and creams, and green tea preparations during the study within the treatment area. Sunscreens were allowed, but were not to be applied in the treatment area within approximately 24 hours before a clinical visit with lesion count.
* Women of childbearing potential were only allowed to participate in this study, if they used a highly effective method of contraception and had a negative serum pregnancy test.

Exclusion Criteria:

* Had known hypersensitivity to 5-aminolevulinic acid (ALA).
* Were subjects under immunosuppressive therapy.
* Suffered from porphyria.
* Showed hypersensitivity to porphyrins.
* Suffered from photodermatoses.
* Had inherited or acquired coagulation defects.
* Had received medication with hypericin or systemically acting drugs with phototoxic or photoallergic potential such as psoralens, tetracyclines, nalidixic acid, furosemide, amiodarone, phenothiazines, quinolones, fibrates, or phytotherapy with St. John's wort, arnica, or valerian or topically applied phototoxic substances like tar, pitch, psoralens or some dyes like thiazide, methylene blue, toluidine blue, eosine, Bengal rose, acridine within 8 weeks prior to treatment with study drug and photodynamic therapy (PDT).
* Had evidence of clinically significant, unstable medical conditions such as

  * metastatic tumor or tumor with high probability of metastatic spread
  * cardiovascular (NYHA class III, IV)
  * immunosuppressive
  * hematological, hepatic, renal, neurological, endocrine
  * collagen-vascular
  * gastrointestinal
* Had currently other malignant or benign tumors of the skin within the treatment area (e.g., malignant melanoma, basal cell carcinoma, invasive squamous cell carcinoma).
* Used any topical treatment in the treatment area within 12 weeks before PDT treatment with BF-200 ALA; biopsy taken at the screening visit was allowed.
* Used topical treatment with ALA or MAL (methyl-aminolevulinic acid hydrochloride) outside the treatment area during participation in the study.
* Systemic treatments of one of the following within the designated period before

PDT with BF-200 ALA:

* Interferon - 6 weeks
* Immunomodulators or immunosuppressive therapies - 10 weeks
* Cytotoxic drugs - 6 months
* Investigational drugs - 8 weeks
* Drugs known to have major organ toxicity - 8 weeks
* Corticosteroids (oral or injectable) - 6 weeks
* Inhaled corticosteroids (>1200 µg/day for beclomethasone, or >600 µg/day for fluticasone) - 4 weeks
* Methyl-aminolevulinic acid hydrochloride or ALA - 12 weeks
* Known allergy against polysorbate 80, caprylic/capric acid triglycerides, isopropyl alcohol, disodium phosphate dihydrate, sodium hydroxide, hydrochloric acid, propylene glycol; sodium benzoate.
* Were known to be pregnant or lactating (currently or within the past 3 months).
* Had any dermatological disease in the treatment area or surrounding area that could be exacerbated by treatment with topical ALA or caused difficulty with examination (e.g. psoriasis, eczema).
* Showed cornu cutaneum like alterations of the skin in the face or on the bald scalp (target area).
* Were currently or within the past 8 weeks participating in another clinical study.
* Had active chemical dependency or alcoholism as assessed by the investigator.
* Confirmed diagnosis of HIV.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof Dr, Principal Investigator — Klinikum der Universität Regensburg Klinik und Poliklinik für Dermatologie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Szeimies RM, Radny P, Sebastian M, Borrosch F, Dirschka T, Krahn-Senftleben G, Reich K, Pabst G, Voss D, Foguet M, Gahlmann R, Lubbert H, Reinhold U. Photodynamic therapy with BF-200 ALA for the treatment of actinic keratosis: results of a prospective, randomized, double-blind, placebo-controlled phase III study. Br J Dermatol. 2010 Aug;163(2):386-94. doi: 10.1111/j.1365-2133.2010.09873.x. Epub 2010 May 28. PMID 20518784
- [Result] Dirschka T, Radny P, Dominicus R, Mensing H, Bruning H, Jenne L, Karl L, Sebastian M, Oster-Schmidt C, Klovekorn W, Reinhold U, Tanner M, Grone D, Deichmann M, Simon M, Hubinger F, Hofbauer G, Krahn-Senftleben G, Borrosch F, Reich K, Berking C, Wolf P, Lehmann P, Moers-Carpi M, Honigsmann H, Wernicke-Panten K, Hahn S, Pabst G, Voss D, Foguet M, Schmitz B, Lubbert H, Szeimies RM; AK-CT002 Study Group; AK-CT003 Study Group. Long-term (6 and 12 months) follow-up of two prospective, randomized, controlled phase III trials of photodynamic therapy with BF-200 ALA and methyl aminolaevulinate for the treatment of actinic keratosis. Br J Dermatol. 2013 Apr;168(4):825-36. doi: 10.1111/bjd.12158. PMID 23252768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period: December 13, 2007 to October 01, 2008. Patients were recruited at 8 study centers in Germany (hospitals and private practices).
Pre-assignment Details: 128 patients were screened, of whom 122 patients were randomized (41 patients to the vehicle/placebo group, 81 patients to the BF-200 ALA group); 6 patients were screening failures (3 patients refused to participate, 3 patients meet exclusion criteria).
Period: Overall Study
Arm/Group | Vehicle | BF-200 ALA
Started | 41 | 81
Completed | 37 | 77
Not Completed | 4 | 4
Not completed — Refused second PDT or withdraw consent | 4 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline description is given for the FAS (Full Analysis Set). One patient each in the vehicle/placebo groupd and in the BF-200 ALA group dropped out without a post-treatment assessment of the target lesions and thus were not considered for the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | BF-200 ALA | Total
Number analyzed (Participants) | 40 | 80 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 10 | 15
  >=65 years | 35 | 70 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.7) | 70.4 (5.2) | 70.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 31 | 72 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 80 | 120
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 40 | 80 | 120
Maximal severity of AK at baseline [Number; unit: participants]
  mild | 11 | 19 | 30
  moderate | 29 | 61 | 90

OUTCOME MEASURES:

1. Primary Outcome: Total Patient Clearance Rate 12 Weeks After the Last Photodynamic Therapy (PDT)
Description: AK clearance rate, defined as the percentage of subjects with complete remission of all AK lesions in the target area(s) assessed 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
Time Frame: 12 weeks after the last photodynamic therapy (PDT), up to 24 weeks
Population: Full analysis set (FAS), Overall
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
percentage of participants | 12.5 [4.2 to 26.8] | 66.3 [54.8 to 76.4]
Statistical Analysis 1: Comparison: Vehicle vs BF-200 ALA; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — The percentages stated relate to the total number of subjects for the respective week and treatment. Cochran-Mantel-Haenszel Test stratified by center

2. Primary Outcome: Total Patient Clearance Rate 12 Weeks After the Last Photodynamic Therapy (PDT)
Description: as for outcome 1
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: per protocol population (PPP), (Overall)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 37 | 77
percentage of participants | 10.8 [3.0 to 25.4] | 63.6 [51.9 to 74.3]
Statistical Analysis 1: Comparison: Vehicle vs BF-200 ALA; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Primary Outcome: Total Patient Clearance Rate Treated With Narrow Spectrum Lamp 12 Weeks After the Last Photodynamic Therapy (PDT)
Description: AK clearance rate, defined as the percentage of subjects with complete remission of all AK lesions in the target area(s) assessed 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
  Analysis was for the subgroup: treated by narrow spectrum lamps only [n=15 (vehicle), n= 31 (BF-200 ALA)]
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS; subgroup analysis for patients only treated with narrow spectrum lamps
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 15 | 31
percentage of participants | 13.3 [1.7 to 40.5] | 87.1 [70.2 to 96.4]

4. Primary Outcome: Total Patient Clearance Rate Treated With Narrow Spectrum Lamp 12 Weeks After the Last Photodynamic Therapy (PDT)
Description: AK clearance rate, defined as the percentage of subjects with complete remission of all AK lesions in the target area(s) assessed 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
  Analysis was for the subgroup: treated by narrow spectrum lamps only [n=13 (vehicle), n= 28 (BF-200 ALA)]
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: PPP; subgroup analysis for patients only treated with narrow spectrum lamps
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 13 | 28
percentage of patients | 15.4 [1.9 to 45.4] | 96.4 [81.7 to 99.9]

5. Secondary Outcome: Percentage of AK Lesions Showing Complete Remission 12 Weeks After the Last PDT
Description: Percentage of individual lesions completely cleared and with no adherent scaling plaques of AK that were visible any longer 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment); Overall population
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS (Overall)
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: individual lesions
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
Number analyzed (individual lesions) | 220 | 455
percentage of lesions | 20.9 [15.7 to 26.9] | 81.1 [77.2 to 84.6]

6. Secondary Outcome: Percentage of AK Lesions Showing Complete Remission Treated With Narrow Spectrum Lamp 12 Weeks After the Last PDT
Description: Percentage of individual lesions completely cleared and with no adherent scaling plaques of AK that were visible any longer 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
  for subgroup analysis: patients treated with narrow spectrum lamp only.
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS, subgroup: lesions treated with narrow spectrum lamp only
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions -PDT with narrow spectrum lamp
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 15 | 31
Number analyzed (lesions -PDT with narrow spectrum lamp) | 86 | 187
percentage of lesions | 15.1 [8.3 to 24.5] | 96.3 [92.4 to 98.5]

7. Secondary Outcome: Change in Total Lesion Size 12 Weeks After the Last PDT
Description: Change in the mean total lesion area 12 weeks per subject after the last PDT compared to baseline (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
  The outcome measure describes the mean difference between total lesion size at baseline and 12 weeks after the last PDT. Negative values indicate a reduction in the total lesion area size compared to baseline.
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS (Overall)
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
mm² | -110.3 (207.9) | -360.2 (194.5)

8. Secondary Outcome: Change in Total Lesion Area 12 Weeks After the Last PDT (Treated Area Face)
Description: Change in mean total lesion area within the target treatment area per subject 12 weeks after the last PDT compared to baseline (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment). The outcome measure describes the mean difference between total lesion size at baseline and 12 weeks after the last PDT. Negative values indicate a reduction in the total lesion area size compared to baseline.
  Subgroup Analysis for patients with lesions located in the face only.
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 29 | 58
mm² | -94.1 (213.0) | -315.0 (198.9)

9. Secondary Outcome: Change in Total Lesion Area 12 Weeks After the Last PDT (Treated Area Scalp)
Description: Change in mean total lesion area within the target treatment area per subject 12 weeks after the last PDT compared to baseline (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment). The outcome measure describes the mean difference between total lesion size at baseline and 12 weeks after the last PDT. Negative values indicate a reduction in the total lesion area size compared to baseline.
  Subgroup Analysis for patients with lesions located in the scalp only.
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mm²
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 15 | 31
mm² | -112.3 (154.5) | -340.2 (194.5)

10. Secondary Outcome: Subjects With Complete Clearance 12 Weeks After the First PDT
Description: AK clearance rate, defined as the number of subjects with complete remission of all AK lesions assessed at 12 weeks after the first PDT
Time Frame: 12 weeks after the first PDT
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
percentage of patients | 10.0 [2.8 to 23.7] | 47.5 [36.2 to 59.0]
Statistical Analysis 1: Comparison: Vehicle vs BF-200 ALA; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

11. Secondary Outcome: Subjects With Partial Clearance 12 Weeks After the Last PDT
Description: Percentage of subjects with clearance of at least 75% of lesions 12 weeks after the last PDT (12 weeks after the 1st PDT or 12 weeks after the 2nd PDT in case of retreatment).
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
percentage of patients | 17.5 [7.3 to 32.8] | 78.8 [68.2 to 87.1]
Statistical Analysis 1: Comparison: Vehicle; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

12. Secondary Outcome: Overall Cosmetic Outcome 12 Weeks After the Last PDT
Description: Overall Cosmetic Outcome (CO) 12 weeks after PDT (12 weeks after 1st PDT or 12 weeks after 2nd PDT). The cosmetic outcome at the end-of-study visit was calculated on the basis of skin quality assessment: skin surface, hyperpigmentation, hypopigmentation, mottled/irregular pigmentation, degree of scarring, and atrophy. The CO was rated as very good if the sum score of the previously mentioned ratings (all ratings for each sign added up) has improved by at least 2 points as compared to baseline; the CO was rated as good if the sum score at a given visit has improved by at least 1 point as compared to baseline; the cosmetic outcome is rated as satisfactory if the sum score at a given visit is identical to the one at baseline; the cosmetic outcome is rated as unsatisfactory if the sum score at a given visit has worsened by 1 point compared to baseline, the cosmetic outcome is rated as impaired if the sum score at a given visit has worsened by at least 2 points compared to baseline.
Time Frame: 12 weeks after the last PDT, up to 24 weeks
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 40 | 80
Participants
  very good | 4 | 19
  good | 6 | 19
  satisfactory | 21 | 39
  unsatisfactory | 5 | 2
  impaired | 4 | 1

13. Secondary Outcome: Local Skin Reactions
Description: Local skin reactions observed immediately after illumination by the investigator were documented using different categories (erythema, edema, induration, vesicles, erosion, ulceration, scaling/flanking, scabbing/crusting,weeping/exudates).
Time Frame: during and after PDT [3h - 4 h]
Population: Safety Population, Overall reactions after first and/or second PDT
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 41 | 81
Participants
  erythema | 15 | 72
  edema | 1 | 32
  induration | 0 | 12
  vesicles | 0 | 0
  erosion | 0 | 0
  ulceration | 0 | 0
  scaling/flaking | 0 | 3
  scabbing/crusting | 0 | 2
  weeping/exudate | 0 | 0

14. Secondary Outcome: Discomfort During and After PDT
Description: Local discomfort experienced by the patient after illumination were documented in three categories: itching, burning, pain.
Time Frame: during and after PDT [3h - 4 h]
Population: Safety Population (Overall reactions after first and/or second PDT)
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 41 | 81
Participants
  pain | 4 | 44
  itching | 0 | 23
  burning | 10 | 70

15. Secondary Outcome: Related Adverse Events /AEs)
Description: Related treatment-emerged-adverse events (TEAEs) until 12 weeks after the last PDT (>=5%) TEAEs were reported from the day of the 1st PDT until the end-of-study (clinical part), i.e. 12 weeks after the last PDT (until 12 weeks after the 1st PDT or up to 24 weeks in case a 2nd PDT was applied).
Time Frame: up to 24 weeks after the 1st PDT
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | BF-200 ALA
Number analyzed (Participants) | 41 | 81
Participants
  Application site erythema | 15 | 72
  Application site irritation | 10 | 70
  Application site pain | 4 | 44
  Application site oedema | 1 | 32
  Application site pruritus | 0 | 27
  Application site induration | 0 | 12
  Application site reaction | 2 | 9

ADVERSE EVENTS:
Time Frame: up to 12 weeks after last treatment (PDT), i.e. 12 weeks after the first PDT or 12 weeks after the second PDT in case of retreatment
Arm/Group | Vehicle | BF-200 ALA
Serious Adverse Events (participants affected / at risk) | 2/41 | 0/81
Other Adverse Events (participants affected / at risk) | 20/41 | 78/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=41) | BF-200 ALA (N=81)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=41) | BF-200 ALA (N=81)
Application site erythema (General disorders) | 15 (22) | 72 (116)
Application site irritation (General disorders) | 10 (11) | 70 (109)
Application site pain (General disorders) | 4 (4) | 44 (62)
Application site oedema (General disorders) | 1 (1) | 32 (39)
Application site pruritus (General disorders) | 0 (0) | 27 (32)
Application site induration (General disorders) | 0 (0) | 12 (14)
Application site reaction (General disorders) | 2 (2) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A publication or presentation of the study results may be planned and initiated by everybody of the scientific personnel involved in this clinical trial but not before the integrated report has been issued. Each party generating the manuscript for publication should allow the other parties a sufficient time in which to review and comment upon the prepublication manuscript.